CLINICAL TRIAL: NCT05424185
Title: Rate of EMG Rise and Rate of Force Development of Scapular Muscles in Overhead Athletes With Different Types of Scapular Dyskinesis
Brief Title: Rate of EMG Rise and Rate of Force Development of Scapular Muscles
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201029RINB
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Scapular Dyskinesis
Keywords: overhead athletes; electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- type 1 scapular dyskinesis: type 1 scapular dyskinesis classified by dyskinesis classification test
  Interventions: Behavioral: different type of scapular dyskinesis
- type 2 scapular dyskinesis: type 2 scapular dyskinesis classified by dyskinesis classification test
  Interventions: Behavioral: different type of scapular dyskinesis
- type 3 scapular dyskinesis: type 3 scapular dyskinesis classified by dyskinesis classification test
  Interventions: Behavioral: different type of scapular dyskinesis
- type 4 scapular dyskinesis: type 4 scapular dyskinesis classified by dyskinesis classification test
  Interventions: Behavioral: different type of scapular dyskinesis

INTERVENTIONS:
Behavioral: different type of scapular dyskinesis — rapid arm elevation to see the different of EMG rise and force development

SUMMARY:
The investigators will clarify rate of electromyography (EMG) rise and rate of force development in overhead athletes on scapular muscles, including upper trapezius, lower trapezius and serratus anterior. The correlation between rate of EMG rise and rate of force development will also be examined.

DETAILED DESCRIPTION:
The contributing factor of scapular dyskinesis can be bony and joint-related issues, neurologic problems, soft tissue problems. Patient with thoracic kyphosis, pectoralis minor stiffness, long thoracic nerve injury, and so on can lead to scapular dyskinesis and further shoulder dysfunction. During shoulder movement, the neuromuscular control of the scapular muscles also play an important role. Previous studies found that participants with pattern 1 and 2 scapular dyskinesis had lesser lower trapezius (5%, P =.025) and serratus anterior activity (10%, P =.004), and higher upper trapezius activity (14%, P =.01) in pattern 2 participants during arm lowering compared to normal participants. Furthermore, the intervention focus on neuromuscular control can change the recruitment pattern of participants with scapular dyskinesis. Significant increases in activation of the middle and lower trapezius (MT: 4.9 ± 2.4% of the maximal voluntary isometric contraction (MVIC); LT: 10.2 ± 6.8% MVIC, p < 0.0 25) were found with conscious control in 3 exercises among the 3 dyskinesis groups, and increased serratus anterior activation (11.2 ± 4.8% MVIC, p < 0.0 25) was found in the concentric phase of side-lying external rotation in the pattern 1 and 1 + 2 groups. The studies show that the muscle recruitment is highly related to the scapular dyskinesis.

However, there are some limitation in the previous studies which presented the outcome by EMG amplitude. First, no matter with or without intervention, previous studies fail to show difference between groups in some condition. Although, there are some difference in lowering phase, the results fail to show difference in elevation phase and some degree of lowering phase. Second, substantial cancellation of the EMG interference signal can occur. The positive and negative signal will be offset. Last, not only neural effect but also contractile effect will be captured. Contraction type, including concentric, eccentric or isometric, will occur in a movement, so the signal will be affected. As the result, another method to represent neuromuscular effect should be considered.

The rate of EMG rise (RER; Formula: ΔEMG/Δtime) has been used to evaluate the rate of muscle activation in order to account for the neural factors that contribute to rate of force development (RFD; Formula: Δforce/Δtime). The onset (<75 ms) of a rapid contraction indicates a role for neural factors. Previous studies with RER outcome have been conducted to see the effect of pain, aging or training. It has been reported that RER reduce with pain and aging while increase after training, and better sensitivity to distinguish difference than peak EMG amplitude (PEMG). The significant difference is found in both upper trapezius and deltoid for RER but only in upper trapezius for PEMG. However, most of the studies about RER are conducted on lower extremity or female worker and no study conducted on athletes, not to mention athletes with scapular dyskinesis.

The overhead sports are characterized with forced and rapid movement. The more sensitive and functional measurement of RER may detect the difference of overhead athletes with different type scapular dyskinesis. Therefore, the purposes of this study are to compare the RER, PEMG, RFD and peak force on scapular muscles (UT, LT, SA) among different types of scapular dyskinesis at 2 arm elevation angles (30, 90 degree). Additionally, to investigate the correlation between RER and RFD. The investigators hypothesize that overhead athletes with scapular dyskinesis will demonstrate significant lower RER and RFD, and there will be significant positive correlation between RER and RFD.

ELIGIBILITY:
Inclusion Criteria:

* Playing overhead sports for at least 1 year.
* Still active in training or competition.
* The frequency of training or game should be at least 2 times per week, 1 hour per time.

Exclusion Criteria:

* Subjects with shoulder pain onset due to trauma, a history of shoulder fractures or dislocation, cervical radiculopathy, degenerative joint disease of the shoulder, surgical interventions on the shoulder, or inflammatory arthropathy.
* Visual analog scale (VAS) > 5 during movement in the experiment.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Scapular dyskinesis is defined as abnormal scapular position and motion. It can be divided in 4 patterns. It has been reported that overhead athletes have higher prevalence (61%) compare to non-overhead athletes (33%). Additionally, athletes with scapular dyskinesis have 43% greater risk of developing shoulder pain than those without scapular dyskinesis. Due to higher prevalence with greater injury risk, scapular dyskinesis plays the important role of injury process that need to be concerned for the overhead athletes.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of EMG rise | Baseline
  Surface EMG electrodes (The Ludlow Company LP, Chocopee, MA) were placed after shaving and preparation with alcohol to decrease skin impedance (typically 10 kΩ or less). An impedance meter (Model F-EZM5, Astro-Med Inc., Ri, USA) will be used to measure impedance between the electrodes and skin over the muscle. Bipolar surface EMG electrodes with an interelectrode (center-to-center) distance of 20 mm will be placed upper trapezius, lower trapezius and serratus anterior of the dominant shoulder. Electrodes for upper trapezius were placed midway between acromion and the seventh spinous process of cervical vertebrae. The lower trapezius was palpated obliquely upward and laterally along the line between intersection of the spine of scapula and the seventh spinous process of thoracic vertebrae. Electrodes for serratus anterior was placed anterior to the latissimus dorsi and posterior to pectoralis major. The reference electrode was placed on the ipsilateral clavicle
rate of force development | Baseline
  The force-sensitive measurement system (FlexiForce ELFTM, New Taipei City, Taiwan, R.O.C.) will be used for force detection. It combines three single-point FlexiForce B201 sensors, one handle containing USB-interface electronics, and Windows-compatible software (Figure 2). Three circle sensors (diameter 9.53 mm; thickness 0.203 mm) are able to detect therange of force as low (4.4-111N), medium (111-667N) and, high level (667-4448N), respectively. This ensures that the various force during measurement can be measured by the appropriate sensor. When the sensor detects the force, the software will display the histogram, curve graph, or number of the force detected as the real-time bio-feedback. The sampling rate of the data collection is set at 200Hz.

SECONDARY OUTCOMES:
Posterior displacement of the scapula | Baseline
  The modified scapulometer will be stationed at one side to measure the distance from the root of the spine (ROS) and the inferior angle (INF) of the scapula to the thoracic wall, respectively. Before conducting the test, two anatomic landmarks, ROS and INF, will be identified and marked. Then two parallel landmarks on the same level of the ROS and INF, approximately 1 cm medial to the scapular medial border, will be marked. The first rater slides the digital caliper anteriorly toward the parallel landmark until firm contact. Posterior displacement of the scapula will be recorded by the second rater based on the digital caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Jiu-Jenq Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] 1. Kibler WB, Ludewig PM, McClure PW, Michener LA, Bak K, Sciascia AD. Clinical implications of scapular dyskinesis in shoulder injury: the 2013 consensus statement from the 'Scapular Summit'. Br J Sports Med 2013;47:877-85. 2. Huang TS, Huang HY, Wang TG, Tsai YS, Lin JJ. Comprehensive classification test of scapular dyskinesis: A reliability study. Manual therapy 2015;20:427-32. 3. McClure P, Tate AR, Kareha S, Irwin D, Zlupko E. A clinical method for identifying scapular dyskinesis, part 1: reliability. J Athl Train 2009;44:160-4. 4. Burn MB, McCulloch PC, Lintner DM, Liberman SR, Harris JD. Prevalence of Scapular Dyskinesis in Overhead and Nonoverhead Athletes: A Systematic Review. Orthopaedic journal of sports medicine 2016;4:2325967115627608. 5. Hickey D, Solvig V, Cavalheri V, Harrold M, McKenna L. Scapular dyskinesis increases the risk of future shoulder pain by 43% in asymptomatic athletes: a systematic review and meta-analysis. Br J Sports Med 2018;52:102-10. 6. Longo UG, Risi Ambrogioni L, Berton A, Candela V, Massaroni C, Carnevale A, et al. Scapular Dyskinesis: From Basic Science to Ultimate Treatment. Int J Environ Res Public Health 2020;17. 7. Huang TS, Ou HL, Huang CY, Lin JJ. Specific kinematics and associated muscle activation in individuals with scapular dyskinesis. Journal of shoulder and elbow surgery 2015;24:1227-34. 8. Ou HL, Huang TS, Chen YT, Chen WY, Chang YL, Lu TW, et al. Alterations of scapular kinematics and associated muscle activation specific to symptomatic dyskinesis type after conscious control. Manual therapy 2016;26:97-103. 9. Huang TS, Du WY, Wang TG, Tsai YS, Yang JL, Huang CY, et al. Progressive conscious control of scapular orientation with video feedback has improvement in muscle balance ratio in patients with scapular dyskinesis: a randomized controlled trial. Journal of shoulder and elbow surgery 2018;27:1407-14. 10. Lawrence JH, De Luca CJ. Myoelectric signal versus force relationship in different human muscles. Journal of applied physiology: respiratory, environmental and exercise physiology 1983;54:1653-9. 11. Jay K, Schraefel M, Andersen CH, Ebbesen FS, Christiansen DH, Skotte J, et al. Effect of brief daily resistance training on rapid force development in painful neck and shoulder muscles: randomized controlled trial. Clin Physiol Funct Imaging 2013;33:386-92. 12. Andersen LL, Andersen JL, Suetta C, Kjaer M, Søgaard K, Sjøgaard G. Effect of contrasting physical exercise interventions on rapid force capacity of chronically painful muscles. J Appl Physiol (1985) 2009;107:1413-9. 13. Andersen LL, Holtermann A, Jørgensen MB, Sjøgaard G. Rapid muscle activation and force capacity in conditions of chronic musculoskeletal pain. Clin Biomech (Bristol, Avon) 2008;23:1237-42. 14. Andersen LL, Nielsen PK, Søgaard K, Andersen CH, Skotte J, Sjøgaard G. Torque-EMG-velocity relationship in female workers with chronic neck muscle pain. Journal of biomechanics 2008;41:2029-35. 15. Weon JH, Kwon OY, Cynn HS, Lee WH, Kim TH, Yi CH. Real-time visual feedback can be used to activate scapular upward rotators in people with scapular winging: an experimental study. J Physiother 2011;57:101-7. 16. Alberta FG, ElAttrache NS, Bissell S, Mohr K, Browdy J, Yocum L, et al. The development and validation of a functional assessment tool for the upper extremity in the overhead athlete. The American journal of sports medicine 2010;38:903-11. 17. Oh JH, Kim JY, Limpisvasti O, Lee TQ, Song SH, Kwon KB. Cross-cultural adaptation, validity and reliability of the Korean version of the Kerlan-Jobe Orthopedic Clinic shoulder and elbow score. JSES open access 2017;1:39-44.